CLINICAL TRIAL: NCT05297383
Title: Pilot: Combining Fish Oil and Exercise to Improve Obesity-Associated Inflammation
Brief Title: Combining HIIT and n-3 PUFA Supplementation to Reduce Inflammation and Improve Metabolic Health (HIIT&PUFA)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Texas Tech University (Other)
Collaborators: University of Houston (Other); Texas Tech University Health Sciences Center (Other)
Responsible Party: Principal Investigator, Kembra Albracht, Assistant Professor, Texas Tech University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-07195-P
Record Dates: First submitted 2022-03-15; First posted 2022-03-28 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Inflammation; Insulin Resistance; Dyslipidemias; Gut Microbiome
MeSH Terms: conditions — Obesity; Inflammation; Insulin Resistance; Dyslipidemias | interventions — Docosahexaenoic Acids; Safflower Oil; High-Intensity Interval Training; Pliability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- n-3 PUFA and flexibility- Control (Active Comparator): Participants will take 4 grams n-3 PUFA (AlaskOmega®) per day (3000 mg EPA and 1000 mg DHA) for 6 weeks. Alongside supplementation, participants will be instructed to maintain their normal level of physical activity but will participate in a time-matched control consisting of flexibility training (low-intensity exercise) for 6 weeks.
  Interventions: Dietary Supplement: Omega-3 Polyunsaturated Fatty Acid.; Behavioral: Flexibility Training
- Placebo and flexibility- Control (Placebo Comparator): Participants will take Placebo (safflower oil, AlaskOmega®, from Organic Technologies Inc.) will be taken by participants in placebo groups for 6 weeks. Alongside supplementation, participants will be instructed to maintain their normal level of physical activity but will participate in a time-matched control consisting of flexibility training (low-intensity exercise) for 6 weeks.
  Interventions: Dietary Supplement: Safflower Oil; Behavioral: Flexibility Training
- n-3 PUFA and HIIT- Test (Active Comparator): Participants will take 4 grams n-3 PUFA (AlaskOmega®) per day (3000 mg EPA and 1000 mg DHA) for 6 weeks. Alongside supplementation, participants will engage in a 4 x 4 HIIT exercise (4 intervals for 4 min at 85-95% HRmax with 3min active recovery at 50-70% HRmax) program, 3 days/week, for 6 weeks.
  Interventions: Dietary Supplement: Omega-3 Polyunsaturated Fatty Acid.; Behavioral: High-Intensity Interval Training
- Placebo and HIIT- Test (Placebo Comparator): Participants will take Placebo (safflower oil, AlaskOmega®, from Organic Technologies Inc.) will be taken by participants in placebo groups for 6 weeks. Alongside supplementation, participants will engage in a 4 x 4 HIIT exercise (4 intervals for 4 min at 85-95% HRmax with 3min active recovery at 50-70% HRmax) program, 3 days/week, for 6 weeks.
  Interventions: Dietary Supplement: Safflower Oil; Behavioral: High-Intensity Interval Training

INTERVENTIONS:
Dietary Supplement: Omega-3 Polyunsaturated Fatty Acid. — 4 grams n-3 PUFA (AlaskOmega®) per day (3000 mg EPA and 1000 mg DHA).
  Other Names: AlaskOmega
  Arms: n-3 PUFA and HIIT- Test; n-3 PUFA and flexibility- Control
Dietary Supplement: Safflower Oil — 4 grams safflower oil (AlaskOmega®) per day.
  Other Names: Placebo
  Arms: Placebo and HIIT- Test; Placebo and flexibility- Control
Behavioral: High-Intensity Interval Training — A 4 x 4 high-intensity interval training (HIIT) exercise program 3 days/week for 6 weeks. This will include a 3 min warm up at 15% watt max followed by 4 intervals for 4 min at 65% watt max with 3 min active recovery at 15% watt max.
  Other Names: HIIT
  Arms: Placebo and HIIT- Test; n-3 PUFA and HIIT- Test
Behavioral: Flexibility Training — 30 min of stretching 3 days/week for 6 weeks
  Other Names: Flexibility
  Arms: Placebo and flexibility- Control; n-3 PUFA and flexibility- Control

SUMMARY:
The goal of this pilot study is to understand the combined effects of fish oil and exercise in obesity-associated inflammation acutely. The investigators hypothesize that fish oil will improve gut bacteria profiles, which will in turn potentiate the benefits of an exercise program and reduce inflammation and metabolic risk.

DETAILED DESCRIPTION:
Incidence of obesity continues to increase in the United States and worldwide, making its prevention or reduction a public health priority. Nutrition research that can lead to effective prevention strategies is greatly needed. Inflammation is a major underlying cause for obesity, and it is imperative that we understand how anti-inflammatory food sources, such as fish oil, could aid in reducing obesity. Moreover, exercise is effective at reducing systemic inflammation and improving insulin resistance. Both exercise and diet can influence health through changes in the gut microbiome; however, no studies have investigated how together these affect gut microbiome and overall metabolic health. The goal is to understand the combined effects of fish oil and exercise in obesity-associated inflammation. The investigators hypothesize that fish oil will improve gut bacteria profiles, which will in turn potentiate the benefits of an exercise program reduce inflammation and metabolic risk. This study will provide the foundation for development of novel strategies for obesity, inflammation, dyslipidemia and dysglycemia.

Aim 1: Determine combined effects of n-3 PUFA and HIIT on improving metabolic risk:

The investigators will test the hypothesis that n-3 PUFA in addition to HIIT will have beneficial effects on obesity-related markers of inflammation, dyslipidemia and insulin resistance in placebo, n-3 or exercise alone, and combined n-3 and exercise.

Aim 1.1: Investigate the influence of n-3 PUFA and HIIT on body weight and composition:

At baseline (week 0), anthropometric assessments will be performed, including: (1) height (m); (2) weight (kg); (3) waist circumference (cm); (4) hip circumference (cm); and body composition which will be assessed utilizing dual-energy X-ray absorptiometry (DXA) scanning. Anthropometric measures will be repeated at post-intervention (week 6).

Aim 1.2: Investigate the influence of n-3 PUFA and HIIT on serum markers associated with obesity

Fasting blood samples collected at weeks 1 and 6 will be analyzed for (1) markers of inflammation, including high sensitivity C-reactive protein (hs-CRP), IL-6, IL-10, MCP-1, and TNF-α; (2) adipokines, including adiponectin, resistin, and leptin; and (3) indices of systemic insulin resistance, including insulin and fasting blood glucose and (4) indices of dyslipidemia, including total cholesterol, high-density, lipoprotein (HDL), non-HDL, low- and very low-density lipoproteins (LDL and VLDL), total/HDL cholesterol, and triglycerides (TG) utilizing ELISA kits or Luminex analyzer [1] in the Nutrition, Exercise, & Translational (NExT) Medicine Lab in the Department of Kinesiology & Sport Management, TTU, Lubbock.

Aim 2: Determine combined effects of n-3 PUFA and HIIT on improving gut dysbiosis:

The investigators will test the hypothesis that n-3 PUFA supplementation will improve gut microbiota composition and related metabolites, which will result in reduced inflammation and ameliorate the metabolic response to a HIIT exercise intervention in an overweight population. This will be accomplished by identifying alterations in gut microbiota profiles following n-3 supplementation, HIIT or the interactive effects of both HIIT and n-3 PUFA.

Aim 2.1: Investigate the influence of n-3 PUFA and exercise on gut microbiota composition

Fecal samples will be collected by participants at their convenience in their homes and less than 24 hours prior to visiting the lab. Samples will be brought to the lab at weeks 1 and 6. Samples will be collected at home with investigator prepared kits and will be stored at -80°C until DNA extraction. Metagenomics analyses will be conducted in consultation with our collaborators at the University of Houston.

Aim 2.2: Investigate the influence of n-3 PUFA and exercise on microbiota produced metabolites

Fecal and serum short-chain fatty acid (SCFA)s, including acetate, propionate and butyrate, will be measured as markers of the above gut bacteria changes and in association with changes in serum markers of inflammation, dyslipidemia and dysglycemia. Fecal and serum SCFAs will be measured utilizing gas chromatography. Analyses will be conducted on fasting blood samples collected at baseline and post-intervention.

Participants will be randomly allocated to 1 of 4 treatment groups (n = 120), each balanced for sex, BMI, lipid profile, and dietary intake.

1. placebo (safflower oil, AlaskOmega®) + flexibility (exercise control)
2. n-3 PUFA (4 grams, 3000 mg EPA and 1000 mg DHA, AlaskOmega®) + flexibility training (exercise control)
3. placebo (safflower oil, AlaskOmega®) + HIIT
4. n-3 PUFA + HIIT

The goal is to conduct the study in smaller cohorts, such as 10-15 participants/group (n = 40-60).

4 grams n-3 PUFA (AlaskOmega®) per day (3000 mg EPA and 1000 mg DHA) will be taken by participants in n-3 PUFA groups for 6 weeks

Placebo (safflower oil, AlaskOmega®, from Organic Technologies Inc.) will be taken by participants in placebo groups for 6 weeks

A 4 x 4 HIIT exercise (4 intervals for 4 min at 85-95% HRmax with 3min active recovery at 50-70% HRmax) program, 3 days/week, conducted under virtual investigator supervision and utilizing cycle ergometers (Keiser M3i Indoor Bike) equipment in collaboration with the TTU Department of Kinesiology & Sport Management for 6 weeks.

If not asked to exercise, participants will be instructed to maintain their normal level of physical activity but will participate in time-matched control consisting of flexibility training led by investigators for 6 weeks.

All participants will wear a heart rate monitor (Polar H10) provided by TTU throughout the training (HIIT and control) to monitor exertion level.

Capsules will be administered in a double-blind fashion and will be identical in appearance. To ensure compliance, subjects will be reminded via phone (text message or phone call based on participant preference) to take their capsules and counts will be conducted when they come in for study visits.

At the end of the 6-week study, assessments will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old.
* Overweight/ Obese.
* Elevated Triglycerides.
* Fasting blood glucose < 126 mg/dL

Exclusion Criteria:

* Diagnosed with diabetes, liver disease, or any lower gastrointestinal disease.
* Currently taking blood pressure, diabetes, or lipid lowering medication.
* Received antibiotic treatment within the last 6 months.
* Are pregnant, lactating, have an irregular menstrual cycle, or are menopausal.
* Currently following a structured or formal weight loss program.
* Exercise ≥ 1 time/week or a moderate-high score on the International Physical Activity Questionnaire.
* Currently taking fish oil supplements (within 4 weeks prior to participant randomization) or eat ≥1 fatty fish meal/week.
* Do not have access to a smartphone.
* Feel uncomfortable riding a stationary bike for 30 minutes.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in Serum high-sensitivity C-reactive protein at 6 weeks | Baseline and 6 weeks
  Serum high-sensitivity C-reactive protein (hs-CRP; mg/L)
Mean Change from Baseline in Interleukin (IL)-6 at 6 weeks | Baseline and 6 weeks
  Interleukin (IL)-6 (pg/mL)
Mean Change from Baseline in Interleukin (IL)-10 at 6 weeks | Baseline and 6 weeks
  Interleukin (IL)-10 (pg/mL)
Mean Change from Baseline in Monocyte chemoattractant protein-1 at 6 weeks | Baseline and 6 weeks
  Monocyte chemoattractant protein-1 (MCP-1; pg/mL)
Mean Change from Baseline in Tumor necrosis factor at 6 weeks | Baseline and 6 weeks
  Tumor necrosis factor (TNF)-alpha (pg/mL)
Mean Change from Baseline in High-density lipoprotein (HDL) at 6 weeks | Baseline and 6 weeks
  High-density lipoprotein (HDL) (mg/dL)
Mean Change from Baseline in Non-high-density lipoprotein (Non-HDL) at 6 weeks | Baseline and 6 weeks
  Non-high-density lipoprotein (Non-HDL) (mg/dL)
Mean Change from Baseline in Low-density lipoprotein (LDL) at 6 weeks | Baseline and 6 weeks
  Low-density lipoprotein (LDL) (mg/dL)
Mean Change from Baseline in Very-low-density lipoprotein (VLDL) at 6 weeks | Baseline and 6 weeks
  Very-low-density lipoprotein (VLDL) (mg/dL)
Mean Change from Baseline in Triglycerides at 6 weeks | Baseline and 6 weeks
  Triglycerides (mg/dL).
Mean Change from Baseline in Total/HDL cholesterol at 6 weeks | Baseline and 6 weeks
  Total/HDL cholesterol (mg/dL)
Mean Change from Baseline in Total cholesterol (mg/dL) at 6 weeks | Baseline and 6 weeks
  Total cholesterol (mg/dL)
Mean Change from Baseline in Insulin at 6 weeks | Baseline and 6 weeks
  Insulin (μU/mL)
Mean Change from Baseline in Fasting blood glucose at 6 weeks | Baseline and 6 weeks
  Fasting blood glucose (mg/dL)
Mean Change from Baseline in Skeletal Muscle Mass Percentage at 6 weeks | Baseline and 6 weeks
  Skeletal Muscle Mass Percentage (%SMM): The percent of the body that is composed of skeletal muscle. Like %BF, this number is relative to total mass.
Mean Change from Baseline in Total Body Fat Percentage at 6 weeks | Baseline and 6 weeks
  Total Body Fat Percentage (%BF): The percent of the body that is composed of fat. This will change based on the amount of fat there is as well as the amount of lean mass there is.
Mean Change from Baseline in Cardio Respiratory Fitness at week 0 | Baseline and 6 weeks
  VO2 Max (mL/kg/min)

SECONDARY OUTCOMES:
Mean Change from Baseline in Bacterial Profile at 6 weeks | Baseline and 6 weeks
  Fecal Microbial DNA (16s Sequencing)
Mean Change from Baseline in Serum Acetate Profile at 6 weeks | Baseline and 6 weeks
  Serum Acetate (SCFA: gas chromatography analysis)
Mean Change from Baseline in Propionate Profile at 6 weeks | Baseline and 6 weeks
  Propionate (liquid chromatography tandem mass spectrometry (LC-MS/MS))
Mean Change from Baseline in Butyrate Profile at 6 weeks | Baseline and 6 weeks
  Butyrate (liquid chromatography tandem mass spectrometry (LC-MS/MS))

CONTACTS AND LOCATIONS:
Overall Officials: Kembra KA Albracht-Schulte, Ph.D., Principal Investigator — Texas Tech University

IPD SHARING:
Plan to Share IPD: No